CLINICAL TRIAL: NCT01324661
Title: The Protective Effect of Friendship on Peer Rejection in Overweight and Normal Weight Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Sarah-Jeanne Salvy, Associate Professor, University at Buffalo
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 3857
Record Dates: First submitted 2010-09-08; First posted 2011-03-29 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Social Exclusion; Control
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Individuals who receive the ball during a computerized ball tossing game about the same number of times as the other players in the game.
- Ostracism (Other): Participant would receive the ball of a ball-tossing game once or twice in the beginning and then never again for the duration of the game.
  Interventions: Behavioral: Ostracism

INTERVENTIONS:
Behavioral: Ostracism — Participants would received the ball of a computerized ball-tossing game once or twice in the beginning and then never again for the duration of the game.
  Arms: Ostracism

SUMMARY:
This study examines youth's motivation for food or social rewards after a brief episode of simulated ostracism. The investigators hypothesize that youth who think about a friend after being ostracized will mediate their decision to resort to food, which is typically evidenced in socially isolated overweight youth.

ELIGIBILITY:
Inclusion Criteria:

* General liking for all study foods

Exclusion Criteria:

* Food allergies
* Medical or Psychological disorders

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2009-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Amount of food consumed after playing a computer game | Measured once during this 3-6 month study
  Participants' food consumption after playing a computer game is measured at the end of the study session
The number of points earned for a snack food or social interaction. | Measured once during this 3-6 month study
  Participants' motivation to earn a reward is measured by the number of mouse clicks participants completed to obtain the reward.

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo Division of Behavioral Medicine, Buffalo, New York, United States